CLINICAL TRIAL: NCT04556656
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel Arm, Multicenter Study Evaluating the Efficacy and Safety of Pridopidine in Patients With Early Stage of Huntington Disease
Brief Title: PRidopidine's Outcome On Function in Huntington Disease, PROOF- HD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prilenia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PL101-HD301; 2020-002822-10 (EudraCT Number)
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Huntington Disease
Keywords: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — pridopidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pridopidine (Experimental): 45 mg pridopidine twice daily (BID)
  Interventions: Drug: Pridopidine
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pridopidine — Pridopidine hard gelatin capsule
  Arms: Pridopidine
Drug: Placebo — Pridopidine-matching placebo hard gelatin capsule
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of pridopidine 45mg twice daily (BID) in patients with early stage manifest Huntington Disease (HD).

DETAILED DESCRIPTION:
This is a phase 3, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of pridopidine 45 mg BID in patients with early stage HD.

ELIGIBILITY:
INCLUSION CRITERIA MAIN STUDY

1. Diagnosis of HD based on clinical features and the presence of ≥36 CAG repeats in the huntingtin gene
2. Diagnostic confidence level (DCL) of 4
3. Adult-onset HD with onset of signs and symptoms ≥18 years of age
4. Stage 1 or Stage 2 HD, defined as a UHDRS-TFC score of ≥7, at screening

EXCLUSION CRITERIA

1. Use of pridopidine within 12 months before the baseline visit.
2. Gene therapy at any time
3. Any serious medical condition or clinically significant laboratory, or vital sign abnormality that precludes the patient's safe participation in and completion of the study e.g. significant heart disease within 12 weeks before baseline or history of certain cardiac arrhythmias
4. History of epilepsy or seizures within the last 5 years
5. Pregnant or breastfeeding, or intention to become pregnant during the study

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yael Cohen, Study Director — Prilenia
Locations (58):
- United States (26):
  - Prilenia Investigational Site (Site 061), Davis, California
  - Prilenia Investigational Site (Site 051), San Diego, California
  - Prilenia Investigational Site (Site 343), Englewood, Colorado
  - Prilenia Investigational Site (Site 333), Washington D.C., District of Columbia
  - Prilenia Investigational Site (Site 160), Gainesville, Florida
  - Prilenia Investigational Site (Site 019), Tampa, Florida
  - Prilenia Investigational Site (Site 032), Atlanta, Georgia
  - Prilenia Investigational Site (Site 088), Chicago, Illinois
  - Prilenia Investigational Site (Site 029), Kansas City, Kansas
  - Prilenia Investigational Site (Site 083), Wichita, Kansas
  - Prilenia Investigational Site (Site 087), Louisville, Kentucky
  - Prilenia Investigational Site (Site 028), Baltimore, Maryland
  - Prilenia Investigational Site (Site 017), Boston, Massachusetts
  - Prilenia Investigational Site (Site 076), Boston, Massachusetts
  - Prilenia Investigational Site (Site 027), St Louis, Missouri
  - Prilenia Investigational Site (Site 037), Albany, New York
  - Prilenia Investigational Site (Site 002), New York, New York
  - Prilenia Investigational Site (Site 119), Durham, North Carolina
  - Prilenia Investigational Site (Site 089), Cincinnati, Ohio
  - Prilenia Investigational Site (Site 020), Columbus, Ohio
  - Prilenia Investigational Site (Site 006), Portland, Oregon
  - Prilenia Investigational Site (Site 018), Philadelphia, Pennsylvania
  - Prilenia Investigational Site (Site 031), Nashville, Tennessee
  - Prilenia Investigational Site (Site 199), Houston, Texas
  - Prilenia Investigational Site (Site 326), Richmond, Virginia
  - Prilenia Investigational Site (Site 096), Seattle, Washington
- Prilenia Investigational site (Site 291), Innsbruck, Austria
- Canada (4):
  - Prilenia Investigational Site (Site 030), Calgary, Alberta
  - Prilenia Investigational Site (Site 048), Vancouver, British Columbia
  - Prilenia Investigational Site (Site 098), Montreal, Quebec
  - Prilenia Investigational Site (Site 232), Halifax
- Prilenia Investigational Site (Site 388), Prague, Czechia
- France (3):
  - Prilenia Investigational Site (Site 385), Lille
  - Prilenia Investigational Site (Site 384), Marseille
  - Prilenia Investigational Site (Site 392), Paris
- Germany (6):
  - Prilenia Investigational Site (Site 234), Aachen
  - Prilenia Investigational Site (Site 379), Bochum
  - Prilenia Investigational Site (Site 377), Lübeck
  - Prilenia Investigational Site (Site 376), Münster
  - Prilenia Investigational site (Site 292), Taufkirchen
  - Prilenia Investigational Site (Site 175), Ulm
- Italy (5):
  - Prilenia Investigational Site (Site 249), Bari
  - Prilenia Investigational Site (Site 394), Bologna
  - Prilenia Investigational Site (Site 239), Milan
  - Prilenia Investigational Site (Site 393), Napoli
  - Prilenia Investigational Site (Site 228), Roma
- Netherlands (2):
  - Prilenia Investigational Site (Site 044), Leiden
  - Prilenia Investigational Site (Site 387), Maastricht
- Poland (3):
  - Prilenia Investigational Site (Site 386), Gdansk
  - Prilenia Investigational Site (Site 244), Krakow
  - Prilenia Investigational Site (Site 246), Warsaw
- Spain (4):
  - Prilenia Investigational Site (Site 380), Barcelona
  - Prilenia Investigational Site (Site 381), Burgos
  - Prilenia Investigational Site (Site 176), Madrid
  - Prilenia Investigational Site (Site 382), Valencia
- United Kingdom (3):
  - Prilenia Investigational Site (Site 180), Aberdeen
  - Prilenia Investigational Site (Site 390), Cardiff
  - Prilenia Investigational Site (Site 378), Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reilmann R, Feigin A, Rosser AE, Kostyk SK, Saft C, Cohen Y, Schuring H, Hand R, Tan AM, Chen K, Feng W, Navon-Perry L, Cruz-Herranz A, Syltevik C, Boot D, Squitieri F, Kayson E, Mehra M, Goldberg YP, Geva M, Hayden MR; PROOF-HD study investigators. Pridopidine in early-stage manifest Huntington's disease: a phase 3 trial. Nat Med. 2025 Nov;31(11):3780-3789. doi: 10.1038/s41591-025-03920-3. Epub 2025 Sep 5. PMID 40913168

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pridopidine | Placebo
Started | 250 | 249
Completed | 222 | 227
Not Completed | 28 | 22
Not completed — Withdrawal by Subject | 14 | 12
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 4 | 7
Not completed — Death | 4 | 0
Not completed — Lost to Follow-up | 3 | 2
Not completed — Not further specified | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pridopidine | Placebo | Total
Number analyzed (Participants) | 250 | 249 | 499
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 207 | 213 | 420
  >=65 years | 43 | 36 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (11.93) | 52.7 (11.39) | 52.5 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 127 | 259
  Male | 118 | 122 | 240
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 2 | 2
  White | 242 | 235 | 477
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 17 | 26
  Austria | 5 | 6 | 11
  Netherlands | 14 | 8 | 22
  United States | 108 | 93 | 201
  Czechia | 6 | 8 | 14
  Poland | 16 | 15 | 31
  Italy | 28 | 30 | 58
  United Kingdom | 5 | 13 | 18
  France | 4 | 7 | 11
  Germany | 37 | 41 | 78
  Spain | 18 | 11 | 29
HD stage at randomization [Count of Participants; unit: Participants]
  HD1 | 102 | 103 | 205
  HD2 | 148 | 146 | 294

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Unified Huntington Disease Rating Scale-Total Functional Capacity (UHDRS-TFC) Score (mITT)
Description: The primary efficacy endpoint for this study was the change from baseline to Week 65 in the TFC (defined as the sum of all TFC 5-items ratings [domestic chores, activities of daily living, finances, care level, and occupation]). The TFC is the standard and well-accepted clinical scale for staging and tracking the progression of HD using functional capacity. Scores range from 0 to 13, with 13 as the least affected and 0 as complete incapacity.
Time Frame: From baseline to Week 65
Population: The modified intent to treat (mITT) population included all participants in the ITT population who received at least one dose of study drug and had valid in clinic TFC scores both at baseline and at least one post-baseline timepoint. The mITT population was analyzed according to the treatment to which the participant was randomized.
  The mITT population was the main analysis population for the primary endpoint in non-EMA regions. Note that the analysis was based on observed data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pridopidine | Placebo
Number analyzed (Participants) | 243 | 247
score on a scale | -1.18 (0.119) | -0.95 (0.119)
Statistical Analysis 1: Comparison: Pridopidine vs Placebo; In the mixed model for repeated measures (MMRM), change from baseline in TFC score was the dependent variable, and independent variables included treatment arm, baseline TFC, region, neuroleptic use or no use, baseline HD stage (HD1 and HD2), categorical week, and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. The unstructured covariance matrix was used for repeated measurements at patient level; Test type: Superiority; p = 0.1670, Mixed Models Analysis; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.54 to 0.09], Standard Error of Mean 0.162

2. Primary Outcome: Change From Baseline to Week 65 in the UHDRS TFC Score (ITT)
Description: as for outcome 1
Time Frame: From baseline to Week 65.
Population: The intent to treat (ITT) population included all randomized participants. The ITT population was analyzed according to the treatment to which the participant was randomized.
  The ITT population was the main analysis population for the primary endpoint in the EMA region.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pridopidine | Placebo
Number analyzed (Participants) | 250 | 249
score on a scale | -1.17 (0.120) | -0.94 (0.120)
Statistical Analysis 1: Comparison: Pridopidine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1598, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.55 to 0.09], Standard Error of Mean 0.162

3. Secondary Outcome: Change From Baseline to Week 65 in Composite UHDRS (cUHDRS) Total Score (mITT)
Description: The composite Unified Huntington Disease Rating Scale (cUHDRS) uses 4 components:
  Total Motor Score (TMS) assesses motor features (oculomotor, dysarthria, chorea, dystonia, gait, postural stability). Higher score = worse outcome. Best score=0. Worst score= 124.
  Stroop Word Reading (SWR) measures attention and mental flexibility. Pat. reads names of colors printed in black ink. Scores reflect correct responses in 45 sec. Higher score = better outcome. Best score=100. Worst score=0.
  Symbol Digit Modalities Test (SDMT) tests psychomotor speed and working memory. Participant has 90 sec to match numbers with symbols. Scores = correct answers in 90 sec. Higher score = better outcome. Best score=120. Worst score=0.
  Total Functional Capacity (TFC) tests the capacity to maintain daily living, finances, care level, occupation. Higher score = better outcome. Best score=13. Worst score=0.
  Total integrated cUHDRS scale range: -7.6 to 24.8. The higher, the better.
Time Frame: From baseline to Week 65
Population: The modified intent to treat (mITT) population included all participants in the ITT population who received at least one dose of study drug and had valid in-clinic TFC scores both at baseline and at least one post-baseline timepoint. The mITT population was analyzed according to the treatment to which the participant was randomized. Note that the analysis was based on as observed data only, patient numbers are therefore lower.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pridopidine | Placebo
Number analyzed (Participants) | 243 | 247
score on a scale | -0.99 (0.109) | -0.88 (0.108)
Statistical Analysis 1: Comparison: Pridopidine vs Placebo; In the MMRM, change in cUHDRS score from baseline was the dependent variable, while independent variables included treatment arm, baseline cUHDRS, region, neuroleptic use or no use, baseline HD stage (HD1 and HD2), categorical week, and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. The unstructured covariance matrix was used for repeated measurements at patient level. No imputation was performed on missing data; Test type: Superiority; p = 0.4544, Mixed Models Analysis; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.4 to 0.18], Standard Error of Mean 0.148

4. Other Pre Specified Outcome: Change From Baseline in cUHDRS Total Score - Patients Off ADMs (mITT)
Description: The composite Unified Huntington Disease Rating Scale (cUHDRS) assesses 4 components (see secondary outcome for details):
  Total Motor Score (TMS) for motor features. Higher score = worse outcome. Worst = 124.
  Stroop Word Reading (SWR) measures attention and mental flexibility. Higher score = better outcome.
  Symbol Digit Modalities Test (SDMT) tests psychomotor speed and working memory. Higher score = better outcome.
  Total Functional Capacity (TFC) tests the capacity to maintain daily living, finances, care level, occupation. The higher, the better.
  Total cUHDRS scale range: -7.6 to 24.8 (assuming 150 as the max score of SWR). The higher, the better.
  This sensitivity analysis was performed in a sub-group of patients who were off neuroleptics AND off vesicular monoamine transporter-2 (VMAT2) inhibitors (together called antidopaminergics, or ADMs) at any time during the study.
Time Frame: Time course from baseline to Week 26, Week 39, Week 52, Week 65, and Week 78
Population: The mITT population was used for subgroup analyses. Note: Analyses/p-values were generated on observed data. Patient numbers at individual weeks varied.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pridopidine | Placebo
Number analyzed (Participants) | 97 | 112
score on a scale
  Week 26: number analyzed (Participants) | 95 | 112
  Week 26 | 0.15 (0.114) | -0.31 (0.108)
  Week 39: number analyzed (Participants) | 90 | 107
  Week 39 | 0.10 (0.130) | -0.34 (0.125)
  Week 52: number analyzed (Participants) | 91 | 104
  Week 52 | -0.07 (0.140) | -0.48 (0.135)
  Week 65: number analyzed (Participants) | 91 | 106
  Week 65 | -0.26 (0.143) | -0.53 (0.137)
  Week 78: number analyzed (Participants) | 70 | 71
  Week 78 | -0.40 (0.159) | -0.54 (0.158)
Statistical Analysis 1: Comparison: Pridopidine vs Placebo; From baseline to Week 26. In the MMRM model, change in cUHDRS score from baseline was the dependent variable and independent variables included treatment group, baseline cUHDRS, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, concomitant use of select medications and Treatment x Concomitant use of select medications, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.0038, Mixed Models Analysis; Mean Difference (Final Values) = 0.46, 95% CI 2-sided [0.15 to 0.76], Standard Error of Mean 0.156
Statistical Analysis 2: Comparison: Pridopidine vs Placebo; From baseline to Week 39; Test type: Superiority; p = 0.0135, Mixed Models Analysis; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [0.09 to 0.80], Standard Error of Mean 0.179
Statistical Analysis 3: Comparison: Pridopidine vs Placebo; From baseline to Week 52; Test type: Superiority; p = 0.0351, Mixed Models Analysis; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [0.03 to 0.79], Standard Error of Mean 0.193
Statistical Analysis 4: Comparison: Pridopidine vs Placebo; From baseline to Week 65; Test type: Superiority; p = 0.1683, Mixed Models Analysis; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.12 to 0.66], Standard Error of Mean 0.197
Statistical Analysis 5: Comparison: Pridopidine vs Placebo; From baseline to Week 78; Test type: Superiority; p = 0.5315, Mixed Models Analysis; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.30 to 0.58], Standard Error of Mean 0.223

5. Other Pre Specified Outcome: Change From Baseline in Q-Motor Finger Tapping Inter-Onset Interval (IOI) Mean - Patients Off ADMs (mITT)
Description: Quantitative (Q)-motor is a clinical assessment of fine motor skills. It is based on the application of pre-calibrated and temperature-controlled force transducers and 3-dimensional position sensors. The index finger is positioned above a force transducer and is to tap as fast as possible. The start was defined as a rise of the force by 0.05 Newton above maximal baseline level. The tap ended when it dropped to 0.05 N before the maximal baseline level was reached again. The IOI refers to the time between the onset of consecutive taps (the faster, the better).
  In addition to the main efficacy analyses, sensitivity analyses were performed in a sub-group of patients who were off neuroleptics AND off vesicular monoamine transporter-2 (VMAT2) inhibitors (together called antidopaminergics, or ADMs) at any time during the study.
Time Frame: Time course from baseline to Week 26, Week 52, Week 65, and Week 78.
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: milliseconds (decrease = improvement)
Arm/Group | Pridopidine | Placebo
Number analyzed (Participants) | 97 | 112
milliseconds (decrease = improvement)
  Week 26: number analyzed (Participants) | 95 | 112
  Week 26 | -14.85 (6.846) | 6.30 (6.449)
  Week 52: number analyzed (Participants) | 91 | 104
  Week 52 | -2.37 (7.135) | 11.95 (6.792)
  Week 65: number analyzed (Participants) | 91 | 104
  Week 65 | -0.79 (7.365) | 23.93 (7.028)
  Week 78: number analyzed (Participants) | 69 | 71
  Week 78 | 1.46 (7.444) | 24.36 (7.230)
Statistical Analysis 1: Comparison: Pridopidine vs Placebo; From baseline to Week 26. In the MMRM model, change in Q-Motor Finger Tapping IOI Mean from baseline was the dependent variable and independent variables included treatment group, baseline Finger Tapping IOI Mean, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, concomitant use of select medications and Treatment x Concomitant use of select medications, with Kenward-Roger approximation for degrees of freedom. No imputation was performed; Test type: Superiority; p = 0.0253, Mixed Models Analysis; Mean Difference (Final Values) = -21.15, 95% CI 2-sided [-39.66 to -2.64], Standard Error of Mean 9.406 — Negative change = improvement
Statistical Analysis 2: Comparison: Pridopidine vs Placebo; From baseline to Week 52; Test type: Superiority; p = 0.1474, Mixed Models Analysis; Mean Difference (Final Values) = -14.31, 95% CI 2-sided [-33.71 to 5.08], Standard Error of Mean 9.853
Statistical Analysis 3: Comparison: Pridopidine vs Placebo; From baseline to Week 65; Test type: Superiority; p = 0.0159, Mixed Models Analysis; Mean Difference (Final Values) = -24.71, 95% CI 2-sided [-44.76 to -4.67], Standard Error of Mean 10.185
Statistical Analysis 4: Comparison: Pridopidine vs Placebo; From baseline to Week 78; Test type: Superiority; p = 0.0283, Mixed Models Analysis; Mean Difference (Final Values) = -22.90, 95% CI 2-sided [-43.34 to -2.45], Standard Error of Mean 10.380

6. Other Pre Specified Outcome: Change From Baseline in Q-Motor Pronation/Supination Inter-Tap-Interval (ITI) Mean - Patients Off ADMs (mITT)
Description: Quantitative (Q)-motor is a clinical assessment of fine motor skills that are crucial for daily activities. It is based on the application of pre-calibrated and temperature-controlled force transducers and 3-dimensional position sensors. Pronation/Supination assesses the regularity of hand taps. The force and duration of the hand taps were recorded similarly to the speeded tapping task. One pronation/supination hand tapping measure is ITI (the faster, the better).
  In addition to the main efficacy analyses, sensitivity analyses were performed in a sub-group of patients who were off neuroleptics AND off vesicular monoamine transporter-2 (VMAT2) inhibitors (together called antidopaminergics, or ADMs) at any time during the study.
Time Frame: Time course from baseline to Week 26, Week 52, Week 65, and Week 78.
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Pridopidine | Placebo
Number analyzed (Participants) | 97 | 112
milliseconds
  Week 26: number analyzed (Participants) | 95 | 112
  Week 26 | -17.63 (8.029) | 20.43 (7.448)
  Week 52: number analyzed (Participants) | 91 | 103
  Week 52 | -0.15 (9.124) | 20.07 (8.555)
  Week 65: number analyzed (Participants) | 91 | 104
  Week 65 | 4.64 (8.380) | 28.55 (7.867)
  Week 78: number analyzed (Participants) | 69 | 70
  Week 78 | 12.73 (9.740) | 34.97 (9.412)
Statistical Analysis 1: Comparison: Pridopidine vs Placebo; From baseline to Week 26. In MMRM model, change in Q-Motor Pronation/Supination ITI Mean from baseline was the dependent variable and independent variables included treatment group, baseline Q-Motor Pronation/Supination ITI Mean, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.0007, Mixed Models Analysis; Mean Difference (Final Values) = -38.06, 95% CI 2-sided [-59.74 to -16.37], Standard Error of Mean 10.999
Statistical Analysis 2: Comparison: Pridopidine vs Placebo; From baseline to Week 52; Test type: Superiority; p = 0.1087, Mixed Models Analysis; Mean Difference (Final Values) = -20.21, 95% CI 2-sided [-44.95 to 4.53], Standard Error of Mean 12.547
Statistical Analysis 3: Comparison: Pridopidine vs Placebo; From baseline to Week 65; Test type: Superiority; p = 0.0395, Mixed Models Analysis; Mean Difference (Final Values) = -23.92, 95% CI 2-sided [-46.68 to -1.16], Standard Error of Mean 11.541
Statistical Analysis 4: Comparison: Pridopidine vs Placebo; From baseline to Week 78; Test type: Superiority; p = 0.1038, Mixed Models Analysis; Mean Difference (Final Values) = -22.23, 95% CI 2-sided [-49.08 to 4.61], Standard Error of Mean 13.587

7. Other Pre Specified Outcome: Change in Q-Motor Pronation/Supination Inter-Onset-Interval (IOI) Mean - Patients Off ADMs (mITT)
Description: Quantitative (Q)-motor is a clinical assessment of fine motor skills that are crucial for daily activities. It is based on the application of pre-calibrated and temperature-controlled force transducers and 3-dimensional position sensors. Pronation/Supination assess the regularity of hand taps. The force and duration of the hand taps were recorded similarly to the speeded tapping task. One pronation/supination hand tapping measure is IOI (the faster, the better).
  In addition to the main efficacy analyses, sensitivity analyses were performed in a sub-group of patients who were off neuroleptics AND off vesicular monoamine transporter-2 (VMAT2) inhibitors (together called antidopaminergics, or ADMs) at any time during the study.
Time Frame: Time course from baseline to Week 26, Week 52, Week 65, and Week 78.
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Pridopidine | Placebo
Number analyzed (Participants) | 97 | 112
milliseconds
  Week 26: number analyzed (Participants) | 95 | 112
  Week 26 | -16.70 (9.399) | 13.68 (8.829)
  Week 52: number analyzed (Participants) | 91 | 103
  Week 52 | 7.40 (10.978) | 24.23 (10.467)
  Week 65: number analyzed (Participants) | 91 | 104
  Week 65 | 7.34 (10.730) | 30.13 (10.232)
  Week 78: number analyzed (Participants) | 69 | 70
  Week 78 | 19.21 (12.702) | 41.93 (12.435)
Statistical Analysis 1: Comparison: Pridopidine vs Placebo; From baseline to Week 26. In the MMRM model, change in Pronation/Supination IOI Mean from BL was the dependent variable and independent variables included treatment group, BL Pronation/Supination IOI Mean, region, categorical week, baseline HD stage (HD1 and HD2), treatment by categorical week interaction, conc. use of select medications and Treatment x Concomitant use of select medications, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.0193, Mixed Models Analysis; Mean Difference (Final Values) = -30.38, 95% CI 2-sided [-55.78 to -4.98], Standard Error of Mean 12.902
Statistical Analysis 2: Comparison: Pridopidine vs Placebo; From baseline to Week 52; Test type: Superiority; p = 0.2680, Mixed Models Analysis; Mean Difference (Final Values) = -16.84, 95% CI 2-sided [-46.69 to 13.02], Standard Error of Mean 15.170
Statistical Analysis 3: Comparison: Pridopidine vs Placebo; From baseline to Week 65; Test type: Superiority; p = 0.1255, Mixed Models Analysis; Mean Difference (Final Values) = -22.79, 95% CI 2-sided [-51.97 to 6.4], Standard Error of Mean 14.829
Statistical Analysis 4: Comparison: Pridopidine vs Placebo; From baseline to Week 78; Test type: Superiority; p = 0.2024, Mixed Models Analysis; Mean Difference (Final Values) = -22.72, 95% CI 2-sided [-57.72 to 12.28], Standard Error of Mean 17.777

8. Other Pre Specified Outcome: Change From Baseline in the UHDRS TFC Score - Patients Off ADMs (mITT)
Description: Total Functional Capacity (TFC) tests the capacity to maintain domestic chores, activities of daily living, finances, care level, and occupation. Scores from 0 - 13. Higher score = better outcome.
  In addition to the main efficacy analyses, sensitivity analyses were performed in a sub-group of patients who were off neuroleptics AND off vesicular monoamine transporter-2 (VMAT2) inhibitors (together called antidopaminergics, or ADMs) at any time during the study.
Time Frame: Time course from baseline to Week 26, Week 39, Week 52, Week 65, and Week 78
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pridopidine | Placebo
Number analyzed (Participants) | 97 | 112
score on a scale
  Week 26: number analyzed (Participants) | 96 | 112
  Week 26 | -0.01 (0.131) | -0.23 (0.124)
  Week 39: number analyzed (Participants) | 92 | 107
  Week 39 | -0.11 (0.137) | -0.31 (0.131)
  Week 52: number analyzed (Participants) | 92 | 106
  Week 52 | -0.19 (0.149) | -0.45 (0.143)
  Week 65: number analyzed (Participants) | 93 | 106
  Week 65 | -0.49 (0.156) | -0.54 (0.150)
  Week 78: number analyzed (Participants) | 71 | 72
  Week 78 | -0.42 (0.166) | -0.54 (0.163)
Statistical Analysis 1: Comparison: Pridopidine vs Placebo; From baseline to Week 26. In the MMRM model, change in UHDRS-TFC score from baseline was the dependent variable and independent variables included treatment group, Baseline UHDRS-TFC, region, categorical week, Baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, concomitant use of select medications and Treatment x Concomitant use of select medications, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.2088, Mixed Models Analysis; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.13 to 0.58], Standard Error of Mean 0.179
Statistical Analysis 2: Comparison: Pridopidine vs Placebo; From baseline to Week 39; Test type: Superiority; p = 0.2991, Mixed Models Analysis; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.17 to 0.57], Standard Error of Mean 0.188
Statistical Analysis 3: Comparison: Pridopidine vs Placebo; From baseline to Week 52; Test type: Superiority; p = 0.2116, Mixed Models Analysis; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-0.15 to 0.66], Standard Error of Mean 0.205
Statistical Analysis 4: Comparison: Pridopidine vs Placebo; From baseline to Week 65; Test type: Superiority; p = 0.8242, Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.38 to 0.47], Standard Error of Mean 0.215
Statistical Analysis 5: Comparison: Pridopidine vs Placebo; From baseline to Week 78; Test type: Superiority; p = 0.5918, Mixed Models Analysis; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.33 to 0.58], Standard Error of Mean 0.231

9. Other Pre Specified Outcome: Change From Baseline in Stroop Word Reading (SWR) - Patients Off ADMs (mITT)
Description: Stroop Word Reading (SWR) measures attention and mental flexibility. Pat. reads names of colors printed in black ink. Scores reflect correct responses in 45 sec. Higher score = better outcome.
  In addition to the main efficacy analyses, sensitivity analyses were performed in a sub-group of patients who were off neuroleptics AND off vesicular monoamine transporter-2 (VMAT2) inhibitors (together called antidopaminergics, or ADMs) at any time during the study.
Time Frame: Time course from baseline to Week 26, Week 39, Week 52, Week 65, and Week 78
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pridopidine | Placebo
Number analyzed (Participants) | 97 | 112
score on a scale
  Week 26: number analyzed (Participants) | 95 | 112
  Week 26 | 2.34 (0.964) | -0.82 (0.916)
  Week 39: number analyzed (Participants) | 91 | 107
  Week 39 | 2.85 (1.100) | -0.04 (1.051)
  Week 52: number analyzed (Participants) | 92 | 104
  Week 52 | 2.73 (1.078) | -0.32 (1.039)
  Week 65: number analyzed (Participants) | 91 | 106
  Week 65 | 1.39 (1.243) | -0.94 (1.193)
  Week 78: number analyzed (Participants) | 70 | 72
  Week 78 | 0.91 (1.261) | -1.08 (1.249)
Statistical Analysis 1: Comparison: Pridopidine vs Placebo; From baseline to Week 26. In the MMRM model, change in SWR score from baseline was the dependent variable and independent variables included treatment group, baseline SWR, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, concomitant use of select medications and Treatment x Concomitant use of select medications, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.0178, Mixed Models Analysis; Mean Difference (Final Values) = 3.16, 95% CI 2-sided [0.55 to 5.77], Standard Error of Mean 1.326
Statistical Analysis 2: Comparison: Pridopidine vs Placebo; From baseline to Week 39; Test type: Superiority; p = 0.0576, Mixed Models Analysis; Mean Difference (Final Values) = 2.89, 95% CI 2-sided [-0.09 to 5.88], Standard Error of Mean 1.518
Statistical Analysis 3: Comparison: Pridopidine vs Placebo; From baseline to Week 52; Test type: Superiority; p = 0.0418, Mixed Models Analysis; Mean Difference (Final Values) = 3.05, 95% CI 2-sided [0.11 to 5.99], Standard Error of Mean 1.493
Statistical Analysis 4: Comparison: Pridopidine vs Placebo; From baseline to Week 65; Test type: Superiority; p = 0.1775, Mixed Models Analysis; Mean Difference (Final Values) = 2.32, 95% CI 2-sided [-1.06 to 5.71], Standard Error of Mean 1.719
Statistical Analysis 5: Comparison: Pridopidine vs Placebo; From baseline to Week 78; Test type: Superiority; p = 0.2627, Mixed Models Analysis; Mean Difference (Final Values) = 1.99, 95% CI 2-sided [-1.50 to 5.48], Standard Error of Mean 1.772

10. Other Pre Specified Outcome: Change From Baseline in Symbol Digit Modalities Test (SDMT) - Patients Off ADMs (mITT)
Description: Symbol Digit Modalities Test (SDMT) tests psychomotor speed and working memory. Participant has 90 sec to write match numbers with symbols. Scoring sums correct substitutions in 90 second interval (max = 110). Higher score = better outcome.
  In addition to the main efficacy analyses, sensitivity analyses were performed in a sub-group of patients who were off neuroleptics AND off vesicular monoamine transporter-2 (VMAT2) inhibitors (together called antidopaminergics, or ADMs) at any time during the study.
Time Frame: Time course from baseline to Week 26, Week 39, Week 52, Week 65, and Week 78.
Population: Note: Analyses/p-values were generated on observed data. Patient numbers at individual weeks varied.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pridopidine | Placebo
Number analyzed (Participants) | 97 | 112
score on a scale
  Week 26: number analyzed (Participants) | 95 | 112
  Week 26 | 0.54 (0.521) | -0.47 (0.484)
  Week 39: number analyzed (Participants) | 91 | 107
  Week 39 | 0.82 (0.512) | -0.06 (0.478)
  Week 52: number analyzed (Participants) | 91 | 104
  Week 52 | -0.42 (0.578) | -0.33 (0.543)
  Week 65: number analyzed (Participants) | 91 | 106
  Week 65 | 0.35 (0.616) | 0.07 (0.576)
  Week 78: number analyzed (Participants) | 70 | 71
  Week 78 | 0.07 (0.617) | -0.36 (0.598)
Statistical Analysis 1: Comparison: Pridopidine vs Placebo; From baseline to Week 26. In the MMRM model, change in SDMT score from baseline was the dependent variable and independent variables included treatment group, baseline SDMT, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.1586, Mixed Models Analysis; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [-0.4 to 2.41], Standard Error of Mean 0.712
Statistical Analysis 2: Comparison: Pridopidine vs Placebo; From baseline to Week 39. In the MMRM model, change in SDMT score from baseline was the dependent variable and independent variables included treatment group, baseline SDMT, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.2144, Mixed Models Analysis; Mean Difference (Final Values) = 0.87, 95% CI 2-sided [-0.51 to 2.25], Standard Error of Mean 0.701
Statistical Analysis 3: Comparison: Pridopidine vs Placebo; From baseline to Week 52. In the MMRM model, change in SDMT score from baseline was the dependent variable and independent variables included treatment group, baseline SDMT, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.9119, Mixed Models Analysis; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-1.65 to 1.48], Standard Error of Mean 0.793
Statistical Analysis 4: Comparison: Pridopidine vs Placebo; From baseline to Week 65. In the MMRM model, change in SDMT score from baseline was the dependent variable and independent variables included treatment group, baseline SDMT, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.7339, Mixed Models Analysis; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-1.38 to 1.95], Standard Error of Mean 0.844
Statistical Analysis 5: Comparison: Pridopidine vs Placebo; From baseline to Week 78. In the MMRM model, change in SDMT score from baseline was the dependent variable and independent variables included treatment group, baseline SDMT, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.6213, Mixed Models Analysis; Mean Difference (Final Values) = 0.43, 95% CI 2-sided [-1.27 to 2.12], Standard Error of Mean 0.859

11. Other Pre Specified Outcome: Change From Baseline in Total Motor Score (TMS) - Patients Off ADMs (mITT)
Description: Total Motor Score (TMS) assesses motor features (oculomotor, dysarthria, chorea, dystonia, gait, postural stability). Each rated 0 (normal) - 4 (abnormal). Higher score = worse outcome. Worst = 124.
  In addition to the main efficacy analyses, sensitivity analyses were performed in a sub-group of patients who were off neuroleptics AND off vesicular monoamine transporter-2 (VMAT2) inhibitors (together called antidopaminergics, or ADMs) at any time during the study.
Time Frame: Time course from baseline to Week 26, Week 39, Week 52, Week 65, and Week 78.
Population: Note: Analyses/p-values were generated on observed data. Patient numbers at individual weeks varied.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pridopidine | Placebo
Number analyzed (Participants) | 97 | 112
score on a scale
  Week 26: number analyzed (Participants) | 96 | 112
  Week 26 | -0.21 (0.568) | -0.03 (0.530)
  Week 39: number analyzed (Participants) | 92 | 107
  Week 39 | 0.06 (0.780) | 0.96 (0.729)
  Week 52: number analyzed (Participants) | 92 | 104
  Week 52 | 0.47 (0.766) | 0.80 (0.720)
  Week 65: number analyzed (Participants) | 91 | 106
  Week 65 | 0.92 (0.847) | 1.28 (0.790)
  Week 78: number analyzed (Participants) | 70 | 72
  Week 78 | 2.19 (0.954) | 1.63 (0.916)
Statistical Analysis 1: Comparison: Pridopidine vs Placebo; From baseline to Week 26. In the MMRM model, change in TMS score from baseline was the dependent variable and independent variables included treatment group, baseline TMS, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.8205, Mixed Models Analysis; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-1.71 to 1.36], Standard Error of Mean 0.777
Statistical Analysis 2: Comparison: Pridopidine vs Placebo; From baseline to Week 39. In the MMRM model, change in TMS score from baseline was the dependent variable and independent variables included treatment group, baseline TMS, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.4028, Mixed Models Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-3.0 to 1.21], Standard Error of Mean 1.067
Statistical Analysis 3: Comparison: Pridopidine vs Placebo; From baseline to Week 52. In the MMRM model, change in TMS score from baseline was the dependent variable and independent variables included treatment group, baseline TMS, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.7577, Mixed Models Analysis; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-2.4 to 1.75], Standard Error of Mean 1.051
Statistical Analysis 4: Comparison: Pridopidine vs Placebo; From baseline to Week 65. In the MMRM model, change in TMS score from baseline was the dependent variable and independent variables included treatment group, baseline TMS, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.7605, Mixed Models Analysis; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-2.64 to 1.93], Standard Error of Mean 1.158
Statistical Analysis 5: Comparison: Pridopidine vs Placebo; From baseline to Week 78. In the MMRM model, change in TMS score from baseline was the dependent variable and independent variables included treatment group, baseline TMS, region, categorical week, baseline HD stage (HD1 and HD2), and treatment by categorical week interaction, with Kenward-Roger approximation for degrees of freedom. No imputation was performed on missing data; Test type: Superiority; p = 0.6694, Mixed Models Analysis; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [-2.05 to 3.18], Standard Error of Mean 1.323

ADVERSE EVENTS:
Time Frame: From Screening until 2 weeks after End of Study/End of Treatment visit (total treatment period of up to 78 weeks).
Arm/Group | Pridopidine | Placebo
All-Cause Mortality (participants affected / at risk) | 4/250 | 1/249
Serious Adverse Events (participants affected / at risk) | 34/250 | 21/249
Other Adverse Events (participants affected / at risk) | 204/250 | 212/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pridopidine (N=250) | Placebo (N=249)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Suicide attempt (Psychiatric disorders) | 3 (3) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal polyp hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (3)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Chorea (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Microcytic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pridopidine (N=250) | Placebo (N=249)
Weight decreased (Investigations) | 13 (13) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 55 (114) | 57 (111)
Contusion (Injury, poisoning and procedural complications) | 12 (20) | 14 (15)
Headache (Nervous system disorders) | 16 (18) | 25 (34)
Diarrhea (Gastrointestinal disorders) | 21 (27) | 22 (32)
Depression (Psychiatric disorders) | 26 (27) | 12 (16)
Anxiety (Psychiatric disorders) | 19 (22) | 16 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 14 (16)
COVID-19 (Infections and infestations) | 59 (62) | 57 (66)
Nasopharyngitis (Infections and infestations) | 19 (22) | 18 (20)
Urinary tract infection (Infections and infestations) | 11 (12) | 17 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs are not employed by the organization sponsoring the study.

There is an agreement between PIs and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

Data and results are owned by the sponsor. Results can be used by the institution for (a) internal noncommercial research, education and patient care, and (b) as required under applicable laws and regulations. Other uses require prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT04556656/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT04556656/SAP_001.pdf